CLINICAL TRIAL: NCT02043873
Title: Can Repair Increase the Useful Life of Composite Resins? Clinical Trial: Triple-blind Controlled - 10 Year Follow-up
Brief Title: Can Repair Increase the Useful Life of Composite Resins?
Acronym: REPCOMP
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Prof. Eduardo Fernández Godoy, University of Chile
Other Study IDs: FOUCH2012/10
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Replacement; Repair; Composites Restorations
Keywords: Clinical Trial; Composite Restorations; Restorations Repair; Replacement Restorations; Operative Dentistry.

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 25 composite restorations replaced: 25 composite replaced with clinically diagnosed secondary caries (Charlie) or undercontoured anatomical form defects (Bravo)
- 25 composite repaired: 25 composite repaired with clinically diagnosed secondary caries (Charlie) or undercontoured anatomical form defects (Bravo)

SUMMARY:
Objectives: The aim of this prospective, randomized, triple-blind cohort study was to assess the longevity of repairs to localized clinical defects in composite restorations that were initially scheduled to be treated with a restoration replacement Methods: 28 patients aged 18 to 80 years with 50 composite restorations were recruited.Restorations with clinically diagnosed secondary caries (Charlie) or undercontoured anatomical form defects (Bravo) were randomly assigned to the Repair (n = 25) or Replacement (n = 25) group, the quality of the restorations was scored according to the modified USPHS criteria. A Wilcoxon test was performed for comparisons between the same groups (CI=0.05). A Friedman test was utilized for multiple comparisons between different years of the same group.

DETAILED DESCRIPTION:
A cohort of 28 patients aged 18 to 80 years of both females (58%) and males (42%) with 50 composite restorations were recruited at the Operative Dentistry Clinic at the Dental School of the University of Chile. All participants presented with one or more clinical features that deviated from the ideal and were rated Bravo or Charlie according to the modified United States Public Health Service (USPHS) criteria 6. The protocol was approved by the Institutional Research Ethics Committee of the Dental School at the University of Chile (Project PRI-ODO-0207). All of the patients signed informed-consent forms and completed a registration form. The selection criteria are summarized below.

2.2 Treatment Group Criteria Initially, 356 restorations (28 patients) were evaluated and assigned in accordance with the modified USPHS criteria, from which 50 were selected in accordance with the inclusion criteria. Restorations with clinically diagnosed secondary caries (Charlie) or undercontoured anatomical form defects (Bravo) were randomly assigned to the Repair (n = 25) or Replacement (n = 25) group (Figure 1). The randomization was performed by the Power Analysis and Sample Size System (PASS software v. 2008, Keysville, UT, USA), and diagnosis of active secondary caries was made based on Ekstrand criteria.

2.3 Restoration Assessment The quality of the restorations was scored according to the modified USPHS criteria. Two examiners underwent calibration exercises each year (JM and EF). The Cohen's Kappa inter-examiner coefficient was 0.74 at the baseline and 0.87 at ten years. Immediately after the treatment (baseline) and 10 years later, the examiners assessed the restorations independently by direct visual and tactile examination with mouth mirror number 5 and explorer number 23 (Hu Friedy Mfg. Co. Inc., Chicago, IL, USA) and indirectly by radiographic examination (bite wing). The five parameters examined were marginal adaptation, anatomic form, surface roughness, secondary caries, and lustre. If a difference was recorded between the two examiners, and if they could not reach an agreement, a third clinician, who also underwent the calibration exercises (GM), made the final decision.

2.4 Treatment Groups 2.4.1 Repair The clinicians (PV - GM) used carbide burs (330-010 Komet, Brasseler GmbH Co., Lemgo, Germany) to explore the defective margins of the restorations, beginning with the removal of part of the restorative material adjacent to the defect to act as an exploratory cavity; this allowed a proper diagnosis and evaluation of the extent of the defect. Provided that the defect was limited and localized, the clinician then removed any defective tooth tissue. Once this material was removed, an exploratory cavity preparation was done that included removal of any demineralized and soft tooth tissue. A self-priming resin bonding system was used (Adper Prompt L-Pop; 3M ESPE, St. Paul, MN, USA), followed by restoration with a resin-based composite (RBC) restorative material (Filtek Supreme; 3M ESPE). A rubber dam isolation was used for this procedure.

2.4.2 Replacement The clinicians totally removed and replaced the defective restorations. After completing the cavity preparations, it was restored with a new resin composite (RC; Filtek Supreme; 3M ESPE). The elimination of the soft tooth tissue caries infection was done using carbide burs at high speed under full water irrigation. During the cavity preparation, no preventive extension or undercutting areas were created, and all of the cavity angles were rounded. In the deep dentin, a glass-ionomer liner was used (Vitrebond; 3M ESPE; USA). Adper Prompt L-Pop, (3M ESPE) was used per the manufacturer instructions, and RBC (Filtek Supreme; 3M ESPE) was applied by the incremental technique. The occlusion was checked, and the restorations were finished and polished following the manufacturer instructions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with localized marginal deficiencies of composite restorations that were clinically judged to be suitable for repair, sealing, or refurbishing according to USPHS criteria (Table 1).
* Patients with more than 20 teeth.
* Restorations in functional occlusions with an opposing natural tooth.
* Asymptomatic restored tooth.
* At least one proximal contact area with a neighbouring tooth.
* Patients older than 18 years.
* Patients who agreed and signed the consent form for participating in the study.
* Area out of the restoration´s failure is in good condition.

Exclusion Criteria:

* Patients with contra-indications for regular dental treatment based on their medical history.
* Patients with special aesthetic requirements that could not be solved by repair treatments.
* Patients with xerostomia or taking medication that significantly decreased salivary flow.
* Patients with a high risk of caries.
* Patients with psychiatric or physical diseases, which interfered with oral hygiene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of 28 patients aged 18 to 80 years (mean 26.5 years) of both females (58%) and males (42%) with 50 composite restorations were recruited at the Operative Dentistry Clinic at the Dental School of the University of Chile
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2003-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Quality composites restorations | up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eduardo Fernández Godoy, Santiango, Met, Chile

REFERENCES:
- [Result] Martin J, Fernandez E, Estay J, Gordan VV, Mjor IA, Moncada G. Management of Class I and Class II Amalgam Restorations with Localized Defects: Five-Year Results. Int J Dent. 2013;2013:450260. doi: 10.1155/2013/450260. Epub 2013 Jan 28. PMID 23431302
- [Result] Martin J, Fernandez E, Estay J, Gordan VV, Mjor IA, Moncada G. Minimal invasive treatment for defective restorations: five-year results using sealants. Oper Dent. 2013 Mar-Apr;38(2):125-33. doi: 10.2341/12-062C. Epub 2012 Jul 11. PMID 22788726
- [Result] Fernandez EM, Martin JA, Angel PA, Mjor IA, Gordan VV, Moncada GA. Survival rate of sealed, refurbished and repaired defective restorations: 4-year follow-up. Braz Dent J. 2011;22(2):134-9. doi: 10.1590/s0103-64402011000200008. PMID 21537587
- [Result] Moncada G, Martin J, Fernandez E, Hempel MC, Mjor IA, Gordan VV. Sealing, refurbishment and repair of Class I and Class II defective restorations: a three-year clinical trial. J Am Dent Assoc. 2009 Apr;140(4):425-32. doi: 10.14219/jada.archive.2009.0191. PMID 19339531
- [Result] Moncada G, Fernandez E, Martin J, Arancibia C, Mjor IA, Gordan VV. Increasing the longevity of restorations by minimal intervention: a two-year clinical trial. Oper Dent. 2008 May-Jun;33(3):258-64. doi: 10.2341/07-113. PMID 18505215
- [Result] Moncada GC, Martin J, Fernandez E, Vildosola PG, Caamano C, Caro MJ, Mjor IA, Gordan VV. Alternative treatments for resin-based composite and amalgam restorations with marginal defects: a 12-month clinical trial. Gen Dent. 2006 Sep-Oct;54(5):314-8. PMID 17004564